CLINICAL TRIAL: NCT04335721
Title: A Pilot Study of Voxelotor for Sickle Cell Anemia Patients at Highest Risk for Progression of Chronic Kidney Disease
Brief Title: A Voxelotor for Sickle Cell Anemia Patients at Highest Risk for Progression of Chronic Kidney Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor voluntarily suspended distribution and removed product from the market
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Global Blood Therapeutics (Industry)
Responsible Party: Principal Investigator, Santosh L Saraf, Principal Investigator, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0047
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Sickle Cell Disease; Sickle Cell Nephropathy
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — voxelotor

STUDY DESIGN:
Intervention Model Description: 6 participants will take voxelotor 1500mg once a day 6 participants will be observed while receiving standard of care (SOC)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Voxelot (Experimental): Voxelotor 1500mg once a day
  Interventions: Drug: Voxelotor
- Standard of Care (SOC) (Other): Observational while receiving SOC
  Interventions: Drug: Voxelotor

INTERVENTIONS:
Drug: Voxelotor — Voxelotor 1500mg once a day

SUMMARY:
This study is a single center, prospective exploratory pilot study of Sickle Cell Anemia (SCA) participants. The study will enroll patients with early stages of sickle cell nephropathy (Chronic Kidney Disease (CKD) stage 1 or 2) who are at the highest risk of CKD progression (presence of both hemoglobinuria and urine albumin concentration ≥ 30 mg/g creatinin

DETAILED DESCRIPTION:
This study is a single center, prospective exploratory pilot study of Sickle Cell Anemia (SCA) participants, age ≥18 years, with SCA. The study will enroll patients with early stages of sickle cell nephropathy (Chronic Kidney Disease (CKD) stage 1 or 2) who are at the highest risk of CKD progression (presence of both hemoglobinuria and urine albumin concentration ≥ 30 mg/g creatinin

ELIGIBILITY:
Inclusion Criteria

1. Documentation of SCA genotype (HbSS or HbSβ0-thalassemia) may be based on history of laboratory testing or must be confirmed by laboratory testing during screening
2. Participants have had urine dipstick defined hemoglobinuria (positive for blood (+1 or higher) and ≤ 2 red blood cells per high power field) on 2 prior outpatient visits
3. Participants with albuminuria (urine albumin ≥ 30 mg/g creatinine) and an eGFR ≥ 60 mL/min/1.73m2 calculated using the CKD-EPI equation on 2 prior outpatient visits
4. Age ≥18 years
5. Hemoglobin (Hb) ≥ 5.5 and ≤ 10.0 g/dL during screening
6. For participants taking hydroxyurea (HU), the dose of HU (mg/kg) must be stable for at least 90 days prior to signing the ICF and with no anticipated need for dose adjustments or initiation during the study, in the opinion of the Investigator
7. Endari stable dose for one month.
8. For participants taking an angiotensin converting enzyme (ACE)-inhibitor or angiotensin receptor blocker, the dose must be stable for at least 90 days prior to signing the ICF and with no anticipated need for dose adjustments or initiation during the study, in the opinion of the Investigator
9. Participants, who if female and of child bearing potential, are using highly effective methods of contraception from study start to 30 days after the last dose of study drug, and who if male are willing to use barrier methods of contraception, from study start to 30 days after the last dose of study drug
10. Participant has provided documented informed consent (the informed consent form [ICF] must be reviewed and signed by each participant

Exclusion Criteria

1. Female who is breast feeding or pregnant
2. Patients who are receiving regularly scheduled blood (RBC) transfusion therapy (also termed chronic, prophylactic, or preventive transfusion) or have received a RBC transfusion for any reason within 30 days of signing the ICF or at any time during the screening period
3. Hospitalized for sickle cell crisis or other vaso-occlusive event within 14 days prior to signing the ICF (i.e., a vaso-occlusive event cannot be within 14 days prior to ICF)
4. Hepatic dysfunction characterized by alanine aminotransferase (ALT) >4 × ULN
5. Participants with clinically significant bacterial, fungal, parasitic or viral infection which require therapy:

   * Participants with acute bacterial infection requiring antibiotic use should delay screening/enrollment until the course of antibiotic therapy has been completed
   * Participants with known active hepatitis A, B, or C or who are known to be human immunodeficiency virus (HIV) positive
6. Severe renal dysfunction (estimated glomerular filtration rate at the Screening visit; calculated by the central laboratory) < 60mL/min/1.732, on chronic dialysis, or have received a kidney transplantation
7. History of malignancy within the past 2 years prior to treatment Day 1 requiring chemotherapy and/or radiation (with the exception of local therapy for non-melanoma skin malignancy)
8. History of unstable or deteriorating cardiac or pulmonary disease within 6 months prior to consent including but not limited to the following:

   * Unstable angina pectoris or myocardial infarction or elective coronary intervention
   * Congestive heart failure requiring hospitalization
   * Uncontrolled clinically significant arrhythmias
9. Any condition affecting drug absorption, such as major surgery involving the stomach or small intestine (prior cholecystectomy is acceptable)
10. Participated in another clinical trial of an investigational agent (or medical device) within 30 days or 5 half-lives of date of informed consent, whichever is longer, or is currently participating in another trial of an investigational agent (or medical device)
11. Inadequate venous access as determined by the investigator/site staff
12. Medical, psychological, or behavioral conditions, which, in the opinion of the Investigator, may preclude safe participation, confound study interpretation, interfere with compliance, or preclude informed consent
13. Receipt of erythropoietin or other hematopoietic growth factors within 28 days of signing ICF or anticipated need for such agents during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Change in albuminuria in voxelotor-treated SCA patients compared to the observation patients by a one-sided test | 48 weeks
  Albuminuria will be analyzed comparing the mean values from the Week 47 and 48 visits to the mean values from the baseline and screening visits

SECONDARY OUTCOMES:
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values in albuminuria | 48 weeks
  Proportion of subjects achieving a 25% decline in albuminuria in the voxelotor-treated group compared to the observation group
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values in kidney function measure | 48 weeks
  24 hour urine protein
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values in In kidney function measure | 48 weeks
  24 hour urine eGFR
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values in kidney function measure | 48 weeks
  24 hour urine albumin concentration
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values in kidney function measure | 48 weeks
  24 hour serum creatinine
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values in Kidney function measure | 48 weeks
  24 hour serum cystatin C
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values in Kidney function measure | 48 weeks
  24 hour serum BUN
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values in Kidney function measure | 48 weeks
  CKD stage
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values kidney function measure | 48 weeks
  24 hour urine retinol binding protein
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values kidney function measure | 48 weeks
  24 hour urine β2 microglobulin
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values kidney function measure | 48 weeks
  Plasma cell-free hemoglobin
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values kidney function measure | 48 weeks
  Urine hemoglobin
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values kidney function measure | 48 weeks
  Urine dipstick-defined hemoglobinuria)
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values markers of hemolysis | 48 weeks
  Lactate dehydrogenase (LDH)
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values markers of hemolysis | 48 weeks
  Aspartate aminotransferase (AST)
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values markers of hemolysis | 48 weeks
  Indirect bilirubin
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values markers of hemolysis | 48 weeks
  Reticulocyte%
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values markers of hemolysis | 48 weeks
  Hemoglobin concentration
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values kidney injury biomarker | 48 weeks
  Urine nephrin
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values kidney injury biomarker | 48 weeks
  Urine podocalyxin
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values kidney injury biomarker | 48weeks
  Urine KIM-1
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values kidney injury biomarker | 48 weeks
  Urine NGAL
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values oxidative injury biomarker | 48weeks
  Serum Methylenedioxyamphetamine (MDA)
Change from the average of the Screening and Baseline values to the Week 47 and Week 48 values oxidative injury biomarker | 48 weeks
  Serum 8-OHd

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois, Chicago, Illinois, United States

REFERENCES:
- [Derived] Obadina M, Wilson S, Derebail VK, Little J. Emerging Therapies and Advances in Sickle Cell Disease with a Focus on Renal Manifestations. Kidney360. 2023 Jul 1;4(7):997-1005. doi: 10.34067/KID.0000000000000162. Epub 2023 May 31. PMID 37254256